CLINICAL TRIAL: NCT05409638
Title: Why am I Still Tired? Adaption, Implementation, and Evaluation of an Intervention for Cancer-Related Fatigue.
Brief Title: Why am I Still Tired ? A Group for Cancer-related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Sophie Lebel, Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 603412-190799-2001
Record Dates: First submitted 2022-05-06; First posted 2022-06-08 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Fatigue; CBT
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT intervention for cancer-related fatigue (Experimental): Participants will receive 4 weekly sessions consisting of psycho-education around fatigue, pacing, journaling fatigue, relaxation training, CBT, and evidence-based tips to increase physical activity.
  Interventions: Behavioral: Cognitive Behavioral Therapy to manage cancer-related fatigue
- Wait-list control group (No Intervention): Participants assigned to this arm wait about 3-months to receive the intervention.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy to manage cancer-related fatigue — Participation will consist of attending 90-minute virtual groups for 4 consecutive weeks on cancer-related fatigue. During the 4 weeks, participants will be asked to participate in activities, participate in group discussions, and complete homework.
  Arms: CBT intervention for cancer-related fatigue

SUMMARY:
Cancer related fatigue (CRF) has been defined as a "distressing, persistent, subjective sense of tiredness or exhaustion related to cancer or cancer treatment that is not proportional to recent activity and interferes with usual functioning". CRF has been found to affect between 59-99% of patients undergoing active treatment. Approximately a third of cancer survivors will continue to experience moderate to severe fatigue upwards of 10 years post-diagnosis. Given the prominence of CRF, guidelines for the assessment and management of CRF have been developed, including guidelines by the Canadian Association for Psychosocial Oncology (CAPO). Despite the availability of guidelines for CRF and a plethora of interventions that have demonstrated effectiveness in aiding patients manage CRF, implementation has been lacking. The objective of this study is to adapt, implement, and evaluate an already existing intervention for CRF in the community using the Knowledge-to-Action framework. This study is an implementation study and evaluation of an evidence-based cognitive-behavioral therapy intervention for CRF in a community setting. An evident knowledge to practice gap exists for CRF management in Ottawa, Canada. Through partnership with a community organization, the Ottawa Regional Cancer Foundation, and an emphasis on long-term sustainability, this project aims to provide more accessible treatment for cancer survivors who are experiencing CRF in the Ottawa region.

DETAILED DESCRIPTION:
This study is a single center, hybrid II effectiveness-implementation pilot study. For the effectiveness trial, the investigators will use a randomized controlled trial with a waitlist control group. For the implementation portion of the study, the investigators will conduct a process evaluation using the RE-AIM framework. Three groups of 10-15 cancer survivors will take part in CrF intervention. Three groups were selected with consultation of the Ottawa Regional Cancer Foundation as it currently offers groups three times a year in the fall, winter, and spring/summer. Another three groups of approximately 10 cancer survivors will be allocated to a 3-month wait-list control group after which they will be offered the CrF intervention. Participants will be recruited through several methods: online advertisements, informational letters and posters sent to community and healthcare organizations and key healthcare providers (i.e., family physicians and health psychologists).

Effectiveness Component:

Participation will consist of attending 90-minute virtual groups for 4 consecutive weeks on cancer-related fatigue. During the 4 weeks, participants will be asked to participate in activities, participate in group discussions, and complete homework. They will also be asked to complete a questionnaire package before the start of the intervention, one week after the intervention is completed (5 weeks), and at 3-months post intervention. The questionnaires package will include the following questionnaires. The primary outcome will be the Multidimensional Fatigue Inventory (MFI-20). Secondary outcomes will be the Functional Assessment of Chronic Illness Therapy (FACIT-F), PROMIS Self-Efficacy for Managing Chronic Conditions-Short Form, Godin Leisure-Time Exercise Questionnaire, The Insomnia Severity Index, and the Hospital Anxiety and Depression Scale (HADS). After the completion of the intervention, they will also be asked to fill out a satisfaction survey once at 5 weeks where they can provide feedback on their experience of the intervention, a component of the process evaluation (see the next section for more detail). All surveys should take approximately 30 minutes. The waitlist control group, participation will consist of completing a 30- minute questionnaire package at the start of the study, after 5 weeks and at a 3-month follow-up. The same questionnaire package will be administered that the intervention group receives with the exception of the satisfaction survey. After three months, participants will be offered the chance to receive the intervention for cancer-related fatigue. They will only be asked to complete the satisfaction survey where they can provide feedback on your experience of the intervention and have the option to participate in the focus group should they wish too. However, they will not be asked to re-complete the questionnaire packages they completed during their wait time. Block randomization with a 1:1 ratio will be completed through an online software. The following sociodemographic data will be collected: age, gender, marital status, education, work class, ethnicity, cancer diagnosis, medication, other chronic illness, history of insomnia and/or depression, smoking, location, income, and comfort with technology.

Implementation component:

This process evaluation will follow a RE-AIM framework. For reach, the investigators will document the number of individuals interested in the intervention and referral sources through the patient demographic form. During past focus groups, the investigators discovered a break-down in communication between community partner, patients, and healthcare organizations. To increase reach and improve this gap, the investigators have several strategies including online advertisements, knowledge dissemination through informational letters to key providers (i.e., family doctors, health psychologists), and offering presenting to community organizations and healthcare organizations. Additionally, feasibility will be assessed retrospectively to examine whether the program was a success or failure, specifically in regard to recruitment, retention, and participation rates. Recruitment numbers and referrals, retention (i.e., percentage of individuals who complete the program), and participation rates (i.e., attendance) will all be tracked throughout the project. If possible, participants will be contacted and asked for the reason of discontinuing the program. For effectiveness, the randomized control trial described above will be conducted. For adoption, the investigators will interview key stakeholders at the Ottawa Regional Cancer Foundation about the barriers and facilitators in maintaining this intervention long-term. The investigators will also be accessing acceptability of the intervention through the evaluation tool created by the Ottawa Regional Cancer Foundation. Evaluation Measure Designed by the Ottawa Regional Cancer Foundation: Currently, programs at the Ottawa Regional Cancer Foundation are routinely evaluated with an evaluation tool. The questionnaire is composed of open-ended questions (e.g., how could the program be improved?) and Likert scales questions on satisfaction (e.g., I would recommend this coaching program to others) and perceived knowledge/skills gained (e.g., this program helped me develop strategies to better cope with life). Further, focus groups (N=3) with 6-10 cancer survivors each who have completed the intervention will be held to gain greater insight into their perspectives of the intervention and which aspects were the most and least beneficial after each group. To assess the quality of training the staff member received, an individual interview will be conducted to ascertain the staff members' confidence and level of preparedness in providing the intervention. In addition, the staff member will be asked about their perspectives of the program and whether they recommend any changes. As the evaluator will be providing the training, the staff interview will be conducted by another graduate student to reduce desirability bias and to ensure the group facilitator can express their honest opinions. For implementation, the investigators will conduct approximate intervention cost-tracking by determining the number of hours the community partner puts into the intervention (i.e., training and facilitating the intervention). Additionally, the intervention will be video recorded, and a fidelity checklist will be completed to ensure high consistency of the intervention. Lastly, for maintenance will be document whether the program is planned to be offered regularly after the investigators have completed our research study

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Has received a cancer diagnosis
* Has completed cancer treatment,
* Self-reports experiencing fatigue,
* Fluent in English.

Exclusion Criteria:

* Currently in treatment
* Has a diagnosis of brain cancer and is experiencing cognitive difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Changes in baseline fatigue at one month | Changes in fatigue at 1 month after the completion of the intervention
  Multidimensional Fatigue Inventory (MFI-20), range from 20 to 100 with higher scores indicating greater fatigue
Changes in baseline fatigue at three months | Changes in fatigue at 3 month after the completion of the intervention
  Multidimensional Fatigue Inventory (MFI-20), range from 20 to 100 with higher scores

SECONDARY OUTCOMES:
Changes in baseline fatigue at 1 month | Changes in fatigue at 1 month after the completion of the intervention
  Functional Assessment of Chronic Illness Therapy (FACIT-F) with a score range 0-52 with higher scores indicating better quality of life and less fatigue
Changes in baseline fatigue at 3 months month | Changes in fatigue at 3 month after the completion of the intervention
  Functional Assessment of Chronic Illness Therapy (FACIT-F) with a score range 0-52 with higher scores indicating better quality of life and less fatigue
Changes in baseline physical activity at 1 month | Changes in physical activity at 1 month after the completion of the intervention
  Godin Leisure-Time Exercise with a score range from 0 to 119 with higher scores indicating greater physical activity
Changes in baseline physical activity at 3 months | Changes in physical activity at 3 month after the completion of the intervention
  Godin Leisure-Time Exercise with a score range from 0 to 119 with higher scores indicating greater physical activity
Changes in baseline depression and anxiety at 1 month | Changes in depression and anxiety 1 month after the completion of the intervention
  Hospital Anxiety and Depression Scale Depression and anxiety (HADS) measure with a range from 0 to 42 with greater scores indicating more distress
Changes in baseline depression and anxiety at 3 months | Changes in depression and anxiety 3 months after the completion of the intervention
  Hospital Anxiety and Depression Scale Depression and anxiety (HADS) measure with a range from 0 to 42 with greater scores indicating more distress
Changes in baseline insomnia at 1 month | Changes in insomnia at 1 month after the completion of the intervention
  Insomnia Severity Index with a score range from 0-28 with higher scores indicating greater insomnia
Changes in baseline insomnia at 3 month | Changes in insomnia at 3 months after the completion of the intervention
  Insomnia Severity Index with a score range from 0-28 with higher scores indicating greater insomnia
Changes in baseline self-efficacy at 1 month | Changes in self-efficacy at 1 month after the completion of the intervention
  PROMIS Self-Efficacy for Managing Chronic Conditions with a score ranging from 0-10 with higher scores indicating greater self-efficacy
Changes in baseline self-efficacy at 3 months | Changes in self-efficacy at 3 months after the completion of the intervention
  PROMIS Self-Efficacy for Managing Chronic Conditions with a score ranging from 0-10 with higher scores indicating greater self-efficacy
Satisfaction with the intervention | One time, 1 month after completing the intervention
  Evaluation Measure Designed by the Ottawa Regional Cancer Foundation with score range from 19 to 95 with higher scores indicating greater satisfaction with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lebel, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No